CLINICAL TRIAL: NCT07245810
Title: Stryker Facial iD Universal Plate Configurator: A Retrospective Post Market Follow Up to Confirm Safety and Performance
Brief Title: Stryker Facial iD Universal Plate Configurator: A Retrospective Post Market Follow Up
Acronym: UPC
Status: Recruiting | Type: Observational
Sponsor: Stryker Craniomaxillofacial (Industry)
Responsible Party: Sponsor
Other Study IDs: UPC_2023_10_CIP_v 1.0
Record Dates: First submitted 2025-08-01; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-08

CONDITIONS: Mandibular Fractures; Facial Fracture; Maxilla Fracture; Orthognathic Surgical Procedures
Keywords: Orthognathic Surgery; Mandibular Reconstruction; Mandibular Fractures; Mandibular Reconstruction* / Methods
MeSH Terms: conditions — Mandibular Fractures; Maxillary Fractures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Orthognatic surgery, Reconstructive maxillofacial surgery, Mandible and maxillofacial trauma surgery — Osteotomy, Mandible and Maxillofacial reconstruction, Orthognathic surgery

SUMMARY:
A retrospective post market follow up to confirm safety and performance of Stryker's Facial iD Universal Plate Configurator (UPC) implants in the clinical setting. The study is performed to confirm the product's performance and safety by systematically collecting clinical data on its use.

DETAILED DESCRIPTION:
This is a retrospective non-interventional post-market follow up aiming at confirming safety and performance of Stryker's Facial iD UPC plating system when used in the clinical setting. This study will include patients who have previously undergone a surgical procedure involving the Study Device, with surgical outcomes evaluated retrospectively. Based on a non-inferiority study power calculation a minimum of 80 patients will be enrolled in the study. Additional patients may be enrolled up to 800 subjects depending on site enrolment rate and patient availability. Up to 3 investigational sites within the United States will participate in this study. The primary outcome parameter evaluating successful fixation or reconstruction of the midface without the need for unplanned revision surgery will be evaluated at all available follow-up timepoints of the included patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who received a Stryker UPC plate for osteotomy, stabilization and rigid fixation of maxillofacial fractures or reconstruction as per routine clinical practice
2. Patients for whom data on the primary outcome variable is available.

Exclusion Criteria:

1. Patients with non-reducible and unstable fractures at the time of surgery
2. Patients with fractures of a severely atrophic mandible at the time of surgery
3. Patients with active local infections at the time of surgery
4. Patients with metal allergies and/or foreign body sensitivity at the time of surgery
5. Patients with limited blood supply or insufficient quality or quantity of bone at the time of surgery
6. Potentially non-compliant patients who are unwilling or incapable of following postoperative care instructions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Eligible patients will be identified as having had a surgical procedure involving the Subject Device.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Successful fixation or reconstruction of the midface without the need for unplanned revision surgery. | Data collected at a single time point per patient in the course of 18 months.
  Assessed by reviewing adverse events in patient medical charts at time point after surgery. Used to document whether an unplanned revision surgery was required or not for patients.

SECONDARY OUTCOMES:
Infection rate | Data collected at time points from patient medical charts in the course of 18 months.
  Determined by adverse events reported from patient medical charts.
Intraoperative complications | Data collected at a single time point per patient in the course of 18 months.
  Determined by adverse events reported from patient medical charts.
Postoperative complications | Data collected at time points per patient in the course of 18 months.
  Determined by adverse events reported from patient medical charts.
Any known adverse events | Data collected at time points per patient in the course of 18 months.
  Determined by adverse events reported from patient medical charts.
Plate failure | Data collected at time points point per patient in the course of 18 months.
  Determined by adverse events reported from patient medical charts.
Satisfactory occlusion achieved after additional orthodontic treatment | Data collected at a single time point per patient in the course of 18 months.
  Data reported in patient medical charts
Time to return to solid food/normal diet | Data collected at a single time point per patient in the course of 18 months.
  Time for patient to return to solid food/normal diet post operation (dd)
Hospitalization time; ICU and normal ward | Data collected at a single time point per patient in the course of 18 months.
  Time the patient was hospitalized post procedure (dd:hh)
EuroQol-5 Domain Questionnaire (if available) | Data collected at time points per patient in the course of 18 months.
  A descriptive system and a visual analogue scale (VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, each with three to five levels of severity. The VAS provides a subjective rating of overall health on a scale from 0 to 100 (higher is better)).
Facial Appearance, Quality of Life, and Satisfaction Questionnaire (if available) | Data collected at time points per patient in the course of 18 months.
  40 independently functioning scales and checklists. Multiple independent scales, each with a 0-100 score, where higher scores indicate better outcomes. Scores are calculated by summing responses on a 4-point Likert scale (e.g., strongly disagree to strongly agree), which are then converted to the 0-100 range. Each scale measures a specific aspect of facial appearance, quality of life, or adverse effects and cannot be summed into a single total score.
12-Item Short Form Health Survey (SF-12) | Data collected at time points per patient in the course of 18 months.
  12 items grouped and scored to produce two separate summary scores: the Physical Component Summary (PCS-12) and the Mental Component Summary (MCS-12). The scale is transformed to a 0-100 range with higher scores indicating better health.

OTHER OUTCOMES:
Primary indication for the surgery / diagnosis | Data collected at a single time point per patient in the course of 18 months.
  Diagnosis collected from patient medical charts.
Max follow-up time | Data collected at a single time point per patient in the course of 18 months.
  Maximum post operative follow up time for patients within standard of care. Reported in patient medical charts during hospital follow up visits.
Surgical approach | Data collected at a single time point per patient in the course of 18 months.
  Surgical approach taken for the procedure. Including: transoral; intraoral; maxillary vestibular approach; transbuccal; submandibular; preauricular; other
Medical conditions | Data collected at time points point per patient in the course of 18 months.
  Underlying medical conditions and medication that may be related to the device or primary outcome.
Localization of the defect | Data collected at a single time point per patient in the course of 18 months.
  Area to treated by the device: mandibular ramus; mandibular body; mandibular condyle; parasymphysis; paramedian; Le Fort I; Le Fort II; Le Fort III; others
Post operative maxillo-mandibular fixation | Data collected at a single time point per patient in the course of 18 months.
  For patients that receive maxillo-mandibular fixation post operation the length of time after surgery the fixation procedure took place (days).
Patient Radiation Exposure | Data collected at time points per patient in the course of 18 months.
  Exposure of patient to radiation therapy within 12 months around the surgery date recorded in patient medical charts (number and type of radiation procedures performed).
  Radiation therapy performed on the anatomical area treated with the device.
  Any postoperative radiation therapy recorded in patient medical charts.
Sterilization method used | Data collected at a single time point per patient in the course of 18 months.
  Sterilization method used for the device. Qualitative responses from site.
Fixation system used | Data collected at a single time point per patient in the course of 18 months.
  System used to fix the device during the procedure. Stryker Universal CMF screws; others
Tightening of screws | Data collected at a single time point per patient in the course of 18 months.
  Tools used to fix the device during the procedure. Response options include :
  Manual and electric screw driver
Orthognathic cases | Data collected at a single time point per patient in the course of 18 months.
  Usage of splints in orthognathic cases.
Year smoking was stopped | Data collected at time points per patient in the course of 18 months.
  Year smoking was stopped (YYYY)
Smoking frequency | Data collected at time points per patient in the course of 18 month
  The frequency of exposure to smoking during periods of smoking (average number of cigarettes per day).
Smoking duration | Data collected at time points per patient in the course of 18 month
  Duration of smoking (pack years)
Years of active smoking | Data collected at time points per patient in the course of 18 month
  Total number of years active smoker (YY)
Patient weight | Data collected at a single time point per patient in the course of 18 months.
  Weight (kg, lb)
Patient height | Data collected at a single time point per patient in the course of 18 months.
  Height (cm, feet, inches)
Patient age | Data collected at a single time point per patient in the course of 18 months.
  Age (years)
Gender | Data collected at a single time point per patient in the course of 18 months
  Responses: Male, Female, undifferentiated, unknown

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - New York Center for Orthognathic and Maxillofacial Surgery, New York, New York
  - New York Center for Orthognathic and Maxillofacial Surgery, Lake Success, New York, New York, New York

REFERENCES:
- See also: Kakarala, Kiran, Yelizaveta Shnayder, Terance T. Tsue, and Douglas A. Girod. 2018. "Mandibular Recon-struction." Oral Oncology. — https://pubmed.ncbi.nlm.nih.gov/29362116/
- See also: Lee, Z. Hye, et al. 2020. "The Latest Evolution in Virtual Surgical Planning: Cus-tomized Reconstruction Plates in Free Fibula Flap M — https://pubmed.ncbi.nlm.nih.gov/32590512/
- See also: Witjes, Max J. H., Rutger H. Schepers, and Joep Kraeima. 2018. "Impact of 3D Virtual Planning on Recon-struction of Mandibular and Maxillary Surgical Defects in Head and Neck Oncology." Current Opinion in Otolaryngology and Head and Neck Surgery. — https://pubmed.ncbi.nlm.nih.gov/29470184/